CLINICAL TRIAL: NCT02927600
Title: Impact of Low Glycemic Responses Breakfast or Dinner on Postprandial Glycemia of the Subsequent Meals
Brief Title: Bed and Breakfast (B&B) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15.18.NRC
Record Dates: First submitted 2016-09-14; First posted 2016-10-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Glycemic response; Glycemic index; Meal intervention; Chinese population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low GI Rice Breakfast (Experimental): Intake of low GI breakfast
  Interventions: Other: Low GI Breakfast
- High GI rice Breakfast (Experimental): Intake of High GI breakfast
  Interventions: Other: High GI Breakfast
- Low GI Rice Dinner (Experimental): Intake of low GI dinner
  Interventions: Other: Low GI Dinner
- High GI Rice Dinner (Experimental): Intake of High GI dinner
  Interventions: Other: High GI Dinner

INTERVENTIONS:
Other: Low GI Breakfast — Intake of low GI breakfast
  Arms: Low GI Rice Breakfast
Other: High GI Breakfast — Intake of high GI breakfast
  Arms: High GI rice Breakfast
Other: Low GI Dinner — Intake of Low GI dinner
  Arms: Low GI Rice Dinner
Other: High GI Dinner — Intake of high GI dinner
  Arms: High GI Rice Dinner

SUMMARY:
The primary objective is to determine which among high vs low Glycemic Index (GI) / Glycemic Responses (GR) interventions at breakfast or at dinner is the most effective for lowering glycemic response of the subsequent standard meal.

DETAILED DESCRIPTION:
Consumption of low Glycemic Index (GI) foods has been shown to not only attenuate blood glucose response during the postprandial period immediately following a meal but to have also positive metabolic effects at the subsequent meal, known as the "second-meal effect" by reducing glucose excursion beyond actual meal. The relative importance of the timing of the glycemic load variation (e.g., breakfast or dinner) on the overall, 24h, glycemic control has not been investigated in detail.

We hypothesize that eating low GI foods in a single meal either for breakfast or for dinner would have different consequential effects on glycemic control over the following meal and thereafter during 24 hours. In order to establish the relative importance of breakfast or dinner in predicting glycemic control/response of the following meal and for a 24-hour period this study will use comprehensive methods including Continuous Glucose Monitoring Systems (CGMS) as well as measuring postprandial blood glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 to ≤ 70 years old years
* Chinese male and female healthy subjects having both grandparents Chinese
* Body mass index: ≥ 18.5 to ≤ 24.9kg/m2
* Waist circumference ≤90 cm for males and ≤ 85 cm for females
* Systolic blood pressure <150 mmHg; Diastolic blood pressure <90 mmHg
* Willing and able to sign written informed consent prior to trial entry

Exclusion Criteria:

* Known Diabetes type 2, under medication
* Fasting Glycemia > 7 mmol/L
* Any clinically relevant gastrointestinal (ulcer, malabsorption), renal (insufficiency), cardiovascular (stroke, arterial hypertension, heart disease), metabolic disease (dyslipidemia), psychiatric disorder (depression) that would affect the study in the opinion of the CNRC clinician, according to a detailed medical history and a blood sampling at screening, only if deemed necessary by CNRC clinician.
* Anemia (anamnesis)
* Subjects who had a history of major gastrointestinal surgery
* Subjects who had more than 5% weight loss from baseline weight during the past three months (more than 5% of initial weight)
* Present drug abuse or use of medications that could interfere with the treatment or energetic metabolism including corticosteroids, growth hormone, hormonal replacement therapy, anti-hypertensives like ACE inhibitor, thiazides and angiotensin receptors blockers. These conditions will be screened based on subject reporting. Participants will be asked to bring in their current medications at the time of screening, and these will be checked by the study-staff.
* Subject allergic /intolerant to any of the test foods or any of the following common food and ingredients: eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings etc.
* Subject on special diets especially vegetarian, high protein or weight loss program.
* Current smokers (i.e. people having smoked in the month preceding the enrolment)
* Subjects having a high alcohol consumption (more than 2 drinks/day)
* Subjects who are not willing and not able to comply with scheduled visits and the requirements of the study procedures in the opinion of the investigators.
* Currently participating or having participated in another clinical trial within 4 weeks prior to trial start.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Glycemia | 3 hours
  Incremental areas under curve (iAUC) of glycemia in the 3 hours following meal intake

SECONDARY OUTCOMES:
Glycemia | 24h
  Incremental areas under curve (iAUC) of glycemia over 24 hours
Plasma glucagon | 3 hours
  Measure of plasma glucagon over a 3-h period following meal intake
Plasma insulin | 3 hours post meal intake
  Measure of plasma insulin over a 3-h period following meal intake
Plasma triglycerides | 3 hours post meal intake
  Measure of plasma triglycerides over a 3-h period following meal intake
Plasma glycerol | 3 hours post meal intake
  Measure of plasma glycerol over a 3-h period following meal intake
Plasma free fatty acids | 3 hours
  Measure of plasma free fatty acids over a 3-h period following meal intake
Satiety | Every 30 minutes over the 3 hours post meal intake
  Satiety will be assessed by Visual Analog Scales
Hunger | Every 30 minutes over the 3 hours post meal intake
  Hunger will be assessed by Visual Analog Scales

CONTACTS AND LOCATIONS:
Overall Officials: Christiani Jeyakumar Henry, Prof, Principal Investigator — Centre for Translational Medicine
Locations (1):
- Clinical Nutrition Research Center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haldar S, Egli L, De Castro CA, Tay SL, Koh MXN, Darimont C, Mace K, Henry CJ. High or low glycemic index (GI) meals at dinner results in greater postprandial glycemia compared with breakfast: a randomized controlled trial. BMJ Open Diabetes Res Care. 2020 Apr;8(1):e001099. doi: 10.1136/bmjdrc-2019-001099. PMID 32327444